CLINICAL TRIAL: NCT02521324
Title: The Effect of Device-Guided Breathing on Healthy Subjects With Sleeplessness Using a Sensor and Mobile App
Brief Title: Effect of Device Guided Breathing on Sleeplessness (2BRT01)
Acronym: 2BRT01
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided to redesign the study.
Sponsor: Afeka, The Tel-Aviv Academic College of Engineering (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2361-15-SMC
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment (IT) (Experimental): Subjects from this group will perform 2 weeks of DGB with the DGB2 system immediately after 1 week of baseline monitoring. All subjects will answer questionnaires pertaining to their sleep quality.
  Interventions: Device: DGB2
- Wait list control (WLC) (Active Comparator): The subjects from the WLC group will do the same (answer questionnaires and perform 2 weeks of DGB with the DGB2 system) at a 1 week delay.
  Interventions: Device: DGB2

INTERVENTIONS:
Device: DGB2 — DGB guides its user in reducing breathing rate gradually from normal values (12-20 breaths/min) to slow rates (4-6 breaths/min) while increasing the relative duration of the exhalation phase. This is done by composing in real time musical tones from monitored respiration data with which the user synchronizes breathing .
  Other Names: Device Guided Breathing

SUMMARY:
The current study is designed to evaluate the effect of device guided breathing (DGB) on sleeplessness. Healthy subjects with mild to moderate sleeplessness that wish to improve their sleep quality will be included in this study. The subjects will receive a belt type breathing sensor, download the app on their smartphone, and will be required to perform DGB at their home setting for 2 weeks after a baseline period.

DETAILED DESCRIPTION:
Sleeplessness, defined as difficulty in falling asleep or maintaining sleep, is prevalent in about one third of the US population. Sleeplessness was found to have negative impact on the quality of life and daily functionality and in its chronic form, was also found to frequently lead to sympathetic over-activity. Stress is an important factor in triggering and exacerbating sleeplessness and its symptoms.

Current methods for alleviating the problem include drugs, modification of sleep habits (also delivered via smartphones), cognitive behavior therapy that includes relaxation techniques such as mindfulness, meditation, and diaphragmatic breathing.

Breathing pattern modification, as done by Device Guided Breathing (DGB) was found to affect beneficially the cardiovascular system. DGB guides its user in reducing breathing rate gradually from normal values (12-20 breaths/min) to slow rates (4-6 breaths/min) while increasing the relative duration of the exhalation phase. This is done by composing in real time musical tones from monitored respiration data with which the user synchronizes breathing

Breathing pattern modification, as done by DGB was originally implemented in a device called RESPeRATE that was cleared by the FDA for treating hypertension and stress and its use was supported by multiple clinical trials. However, the direct effect of DGB on sleeplessness has not yet been investigated,

DGB was recently implemented in a mobile system that consists of a Bluetooth enabled belt-type breathing sensor and an iOS mobile application ('App'). The App accumulates continuously breathing-related data and performance measure. The accumulated data are sent to an icloud-based server.

The current study is a single center, prospective, randomized, waiting-list-controlled (WLC) clinical trial designed to evaluate the effect of DGB on sleeplessness using the mobile DGB2 system.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy with mild to moderate sleeplessness
2. Male or Female, Age 18-65
3. Has ipod/ipad or smartphone compatible with the system used in the study
4. Has access to internet and email
5. Knowledge of English to the level of understanding the App and the sleep-monitor interface.

Exclusion Criteria:

1. Known sleep or respiration disorder
2. A serious systemic disease
3. Pittsburg Insomnia Rating Scale (PIRS_2) <2
4. Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change in Energetic/Fatigue visual analogue scale (VAS) from baseline to completion of 2 weeks of DGB | 2 weeks

SECONDARY OUTCOMES:
Changes in sleep onset latency (SOL) from baseline to completion of 2 weeks of DGB | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Halak, MD, Principal Investigator — Sheba Medical Center; Zehava Blechman, PhD, Study Director — Afeka, Tel-Aviv Academic College of Engineering/
Locations (1):
- Afeka, Tel-Aviv Academic College of Engineering, Tel Aviv, Please Select Region, State Or Province, Israel

IPD SHARING:
Plan to Share IPD: Undecided